CLINICAL TRIAL: NCT06600295
Title: Oncology, Undernutrition and Sensoriality: Links, Mechanisms and Levers for Action - Study ONDES
Brief Title: Oncology, Undernutrition and Sensoriality: Links, Mechanisms and Levers for Action
Acronym: ONDES
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: COTTET INCa SHSESP 2023
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Newly Diagnosed Cancer of the Oropharynx, Oral Cavity, Colon or Liver
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- patients with cancer of the oral cavity/oropharynx: 115 patients with cancer of the oral cavity/oropharynx
  Interventions: Other: tests/questionnaires; Biological: biological samples; Other: evaluation
- colon cancer patients: 123 colon cancer patients
  Interventions: Other: tests/questionnaires; Biological: biological samples; Other: evaluation
- patients with liver cancer: 68 patients with liver cancer
  Interventions: Other: tests/questionnaires; Biological: biological samples; Other: evaluation

INTERVENTIONS:
Other: tests/questionnaires — EVA, LFPQ-fr, Taste strips, ETOC 6-items, CiTAS, Fr-sQOD, WHOQOL-Bref, HADS
Biological: biological samples — blood, saliva, tongue mucus
Other: evaluation — strength tests using handgrip tests, chair lifts or walking speed and sarcopenia tests for the over-70s

SUMMARY:
Cancers of the upper aerodigestive tract account for around 4% of all malignant tumours worldwide. Colon and liver cancer are the most common digestive cancers. The epidemiology of liver cancer is changing, and the number of deaths from liver cancer has increased by 25% worldwide (Huang 2022). In France, around 19,000 cancers of the upper aerodigestive tract and 88,000 new cases of digestive cancer are diagnosed each year (colon cancer remains the most common) (Globocan 2020). Patients with these two types of cancer are at particularly high risk of undernutrition (Pressoir 2010; Gyan 2018).

In cancer patients, changes in diet may result from constraints linked to the cancer or possible after-effects, but also from personal choices (for example, adopting a healthier diet). Cancer and its treatment lead to changes such as increased nutritional requirements and hypercatabolism, or sensory changes (taste and smell), reducing pleasure and food intake. These problems will impair quality of life and intensify undernutrition, a major problem in the management of the disease since it increases the risk of complications, therapeutic failure and mortality. It is estimated that 10-20% of deaths in cancer patients are attributable to the consequences of undernutrition rather than to the disease itself (Pressoir 2010). In the VICAN study, 41% of patients changed their diet after diagnosis: 29% because of changes in taste and 82% to have a healthier diet (INCa 2014). These changes were associated with the treatment received, the presence of sequelae and anxiety.

Taste and smell disorders are common in different types of cancer (any solid or haematological type) and treatments (chemotherapy, radiotherapy and surgery) (De Conno 1989; Heckel 2015; Spotten 2017; van Oort 2018). The mechanisms involved in sensory changes are not fully understood, especially in cancer, and with different types and treatments (Murtaza 2017). Several hypotheses have been proposed: altered expression of enzymes of the oral sphere, altered expression of sensory receptors (Neiers 2021), saliva composition and function (Zhu 2021), and impact of the oral microbiota (Schwartz 2021a, Licandro 2023).

The early identification of undesirable effects linked to nutrition, and the early or anticipated diagnosis of undernutrition are important issues in the management of cancer patients. The pleasure (or displeasure) produced by food guides desire and eating behaviour. The mechanisms involved are linked to hedonic sensations: conditioned satiety, specific sensory satiety, negative alliesthesia and the reward system (hedonic system). The latter is influenced by the environment and can be consciously controlled, with several dimensions: liking (the patient likes or dislikes a given food) and wanting (evaluates the desire to consume a given food at a given moment). All these parameters, together with sensory and dietary learning throughout life (habits, beliefs and constraints), influence food preferences and therefore eating behaviour. Individual sensitivities and the personal history of the disease (treatment and care pathway, sequelae, presence of co-morbidities, etc.) must therefore be taken into account when setting up preventive actions for cancer patients. It seems important to explore these factors, the experience of patients and the consequences for eating behaviour in daily life, in order to improve support and communication with healthcare professionals, as well as prevention and early detection of undernutrition. It would be interesting to conduct more in-depth studies on nutritional status, quality of life and changes in taste and smell, which in most studies have been considered separately.

ELIGIBILITY:
Inclusion Criteria:

Patient :

* With newly diagnosed cancer of the oropharynx, oral cavity, colon or liver (at any stage).
* For whom first-line treatment has been decided including radiotherapy, chemotherapy, immunotherapy and/or surgery.
* Able to follow all study procedures in accordance with the protocol.
* Have given their oral, free and informed consent to participate in the study.

Exclusion Criteria:

* Person not affiliated with national health insurance system
* Person subject to a legal protection measure (curatorship, guardianship)
* Pregnant women, women in labour or breastfeeding mothers
* Adults who is unable to give consent
* Minors
* Person unable to read, speak, write and understand French
* Patients with neuro-cognitive disorders (post-stroke, dyslexia, dyspraxia) or neuro-psychiatric disorders (dementia, autism) that make it impossible to assess taste sensoriality.
* Patients with olfactory or gustatory disorders documented prior to the disease
* Patient with another cancer currently being treated
* Patients with a systemic disease or physical trauma affecting taste perception
* Patients with kidney failure
* Patients with sinonasal polyposis
* Patients undergoing immunosuppressive treatment
* Patients with an estimated life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified :
  * at the department's multidisciplinary consultation meetings
  * during consultations with their referring doctor (ENT or gastroenterologist)
Sampling Method: Non-Probability Sample
Enrollment: 306 (Estimated)
Dates: Start 2024-09-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The presence or absence of undernutrition | Through study completion, an average of 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France